CLINICAL TRIAL: NCT07354256
Title: Acute Effects of Percussive Therapy Intensity on Agility, Vertical Jump Kinetics, and Neuromuscular Performance Across Morning and Evening Sessions in Trained Male Football Players
Brief Title: Acute Effects of Percussive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monira Aldhahi (Other)
Responsible Party: Sponsor-Investigator, Monira Aldhahi, Associate Prof, Princess Nourah Bint Abdulrahman University
Organization: Princess Nourah Bint Abdulrahman University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PNU-9
Record Dates: First submitted 2026-01-07; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Health Adult Subjects
Keywords: vibration therapy; football

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PASSIVE REST (Control) (Other): Participants rested in a seated position for 5 minutes with no massage applied. This condition served as the passive control to account for baseline performance and circadian variation.
  Interventions: Other: Passive Rest
- Low-Intensity Percussive Massage (28 Hz) (Experimental): Participants received low-intensity percussive massage using a handheld massage device at 28 Hz for a total duration of 5 minutes (2.5 minutes per leg), targeting the quadriceps, hamstrings, and gluteal muscles.
  Interventions: Device: Percussive Massage Therapy
- Moderate-Intensity Percussive Massage (35 Hz) (Experimental): Participants received moderate-intensity percussive massage using a handheld massage device at 35 Hz for a total duration of 5 minutes (2.5 minutes per leg), targeting the quadriceps, hamstrings, and gluteal muscles.
  Interventions: Device: Percussive Massage Therapy

INTERVENTIONS:
Device: Percussive Massage Therapy — Percussive massage therapy was delivered using a handheld device (Hypervolt 2 Pro) applied bilaterally to the quadriceps, hamstrings, and gluteal muscles. The total intervention duration was 5 minutes (2.5 minutes per leg). Two intensity levels were used: low intensity at 28 Hz and moderate intensity at 35 Hz. The device was applied using continuous longitudinal strokes at a controlled speed by a trained investigator immediately after a standardized warm-up.
  Arms: Low-Intensity Percussive Massage (28 Hz); Moderate-Intensity Percussive Massage (35 Hz)
Other: Passive Rest — Participants remained seated at rest for 5 minutes with no massage or device application. This condition served as the passive control to account for baseline performance and circadian variation.
  Arms: PASSIVE REST (Control)

SUMMARY:
This randomized crossover study investigates the acute effects of different percussive massage intensities on agility, jumping, strength, and power performance in trained male football players. Participants complete three experimental conditions (no massage, low-intensity percussive massage, and moderate-intensity percussive massage) at two different times of day (morning and evening). Performance outcomes are assessed immediately following each intervention to examine dose-response effects and potential interactions with circadian timing.

ELIGIBILITY:
Inclusion Criteria:

* Male football players aged 18-25 years
* Possession of an active football license
* Minimum of 2 years of systematic football training experience
* Regular participation in football training at least three times per week
* Willingness and ability to attend both morning and evening testing sessions
* Ability to provide written informed consent

Exclusion Criteria:

* Presence of any acute or chronic musculoskeletal injury
* History of neurological disorders
* Any medical condition that could affect neuromuscular performance or limit safe participation
* Current illness, pain, or discomfort during the study period
* Inability to complete all experimental sessions or comply with study procedures

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Agility Performance | Immediately post-intervention (morning and evening sessions)
  Agility performance assessed using the T-Test
  T-Test: A cone configuration was set up forming a "T" shape (10 m forward, 5 m to the left, and 5 m to the right). The participants sprinted forward, shuffled laterally to the left and right, and backpedaled to the starting position.
Countermovement Jump Height | Immediately post-intervention (morning and evening sessions)
  Vertical jump height (cm) measured using the Countermovement Jump test via the My Jump Lab smartphone application. The highest value from three maximal trials was retained for analysis.
  Time Frame:
Agility | Immediately post-intervention (morning and evening sessions)
  Illinois Agility Test: Participants started from a prone position (chest on the floor), stood up, and sprinted through a slalom course marked by cones over a 10 m × 5 m area.
  The timing was recorded to the nearest 0.01 s using electronic timing gates (Brower Timing Systems, Draper, UT, USA). The participants performed two trials for each agility test, and the best performance was retained for statistical analysis.

SECONDARY OUTCOMES:
Vertical jump performance | Immediately post-intervention (morning and evening sessions)
  Vertical jump performance parameters were assessed using the Countermovement Jump (CMJ) test via the My Jump Lab application (v.4.4.2, developed by Dr. Carlos Balsalobre). This smartphone-based application uses high-speed video analysis to calculate jump variables and has been validated against gold-standard force platforms

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University/ PNU, Riyadh, Saudi Arabia, Saudi Arabia